CLINICAL TRIAL: NCT07062003
Title: A Dose Finding Study of MiniBeam RadioTherapy for Skin and Superficial Soft Tissue Tumors (MBRT1)
Brief Title: Minibeam Radiation Therapy With Tungsten Slit Collimator for the Treatment of Recurrent or Metastatic Skin or Soft Tissue Tumors, MBRT1 Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMROR2471; NCI-2025-04429 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-004810 (Other: Mayo Clinic Institutional Review Board); GMROR2471 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Malignant Skin Neoplasm; Metastatic Malignant Soft Tissue Neoplasm; Recurrent Malignant Skin Neoplasm; Recurrent Malignant Soft Tissue Neoplasm; Skin Neoplasm; Soft Tissue Neoplasm
MeSH Terms: conditions — Skin Neoplasms; Sarcoma; Soft Tissue Neoplasms | interventions — Biopsy; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Device feasibility (MBRT with tungsten slit collimator) (Experimental): Patients undergo MBRT with a tungsten slit collimator over 2-3 fractions on study. Patients also undergo standard of care CT simulation on study and undergo collection of blood samples and punch or core biopsy throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Medical Device Usage and Evaluation; Radiation: Minibeam Radiation Therapy

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Other: Medical Device Usage and Evaluation — Undergo MBRT with tungsten slit collimator
Radiation: Minibeam Radiation Therapy — Undergo MBRT with tungsten slit collimator
  Other Names: MBRT

SUMMARY:
This clinical trial tests the safety and best dose of minibeam radiation therapy (MBRT) with a tungsten slit collimator for treating patients with skin or soft tissue tumors that have come back after a period of improvement (recurrent) or that spread from where they first started (primary site) to other places in the body (metastatic). Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill tumor cells and shrink tumors. Tungsten is an extremely dense metal and is commonly used for blocking x-rays for minimum radiation exposure. A tungsten slit collimator is a device that separates an initially wide beam of x-rays into several very narrow individual beams of radiation. As radiation passes through the collimator, the radiation hits regions of solid tungsten and is blocked. In the open slit regions, radiation passes through to the intended target/tumor area defined by the physician. The tungsten slit collimator then selectively blocks portions of the radiation to create an alternating pattern of higher "peak" and lower "valley" radiation dose regions. These narrow beams of radiation are referred to as "minibeams" and the general approach referred to as MBRT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose (MTD) of MBRT and describe the adverse events of treatment.

SECONDARY OBJECTIVE:

I. To assess the ability to maintain a distinct differential between peak and valley doses using film dosimetry.

EXPLORATORY OBJECTIVES:

I. To estimate the rate of freedom from local progression at 6 and 12 months after the start of MBRT.

II. To evaluate pre-treatment and post-treatment differential abundance of peripheral blood immune cell populations and their activation markers.

III. Explore germline and somatic mutations in homologous recombination (HR) genes and their association with freedom from local progression.

IV. Quantify the immune phenotypes and cell signaling in the tumor microenvironment pre-MBRT and post-MBRT using bulk ribonucleic acid (RNA)-sequencing (seq) data.

OUTLINE:

Patients undergo MBRT with a tungsten slit collimator over 2-3 fractions on study. Patients also undergo standard of care CT simulation on study and undergo collection of blood samples and punch or core biopsy throughout the study.

After completion of study treatment, patients are followed up at weeks 2, 4, and 12, and months 6, 9, and 12.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed malignancy
* Primary, recurrent, or metastatic skin or superficial soft tissue tumor amenable to palliative orthovoltage radiotherapy
* Anticipated life expectancy ≥ 30 days and anticipated capacity for follow up for ≥ 30 days
* Negative pregnancy test done ≤ 28 days prior to registration, for biological women of childbearing potential only
* Willing to provide written informed consent
* Willing to allow baseline and follow up photograph acquisition for response and toxicity assessment
* Willing and able to return to enrolling institution for follow-up during the active monitoring phase of the study
* Willing to provide blood and tissue samples for correlative research purposes

Exclusion Criteria:

* Hematologic, germ cell, or any other tumor that the investigational team would deem to have a high likelihood of clinical complete response with standard palliative radiotherapy (8 Gy in 1, 30 Gy in 10, etc.)
* COHORT A (INTACT SKIN) ONLY: Prior radiotherapy targeting the lesion presenting for treatment or prior adjacent radiotherapy if > 10 Gy overlaps with a portion of the planned target
* Treatment with a B-Raf proto-oncogene, serine/threonine kinase (BRAF) inhibitor, monoclonal antibodies targeting vascular endothelial growth factor (VEGF) (bevacizumab or ramucirumab) or small molecule inhibitors inhibiting VEGF within the last 2 weeks or planned treatment with BRAF inhibitor within 4 weeks after radiation
* Treatment with an investigational drug therapy within 2 weeks prior to or 4 weeks (the DLT monitoring period) after MBRT
* Any tumor with direct extension into the spine such that targeting the spine/spinal cord could not be avoided

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | Up to 28 days
  The maximum tolerated dose is defined as the dose level associated with a dose limiting toxicity (DLT) probability closest to the target toxicity rate (30%), which will be determined based on the time-to-event Bayesian optimal interval procedures. The incidence and proportion of patients experiencing DLTs will be summarized for each dose level and across all dose levels.
Incidence of adverse events | Up to 12 months
  Safety will be assessed based on reported adverse events (AEs). The severity of AEs will be graded as mild, moderate, severe, or life-threatening according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Ability to maintain a distinct differential between peak and valley doses using film dosimetry | Up to 12 months
  Film dosimetry will be obtained for every patient treatment. Radiochromic film will be placed directly on the tumor. Will measure and record peak and valley doses as well as the resulting peak-to-valley dose ratio.
Incidence of adverse events | At months 6, 9, and 12
  Safety will be assessed by CTCAE 5.0 by investigating (1) grade 3 AEs deemed possibly, probably, or definitely related to study treatment and (2) all grade 4-5 AEs regardless of attribution to the study treatment. The proportions of patients with these AEs at months 6, 9, and 12 will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Scott C. Lester, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials